CLINICAL TRIAL: NCT01677767
Title: Efficacy of C.E.R.A. for Correction of Anemia and Maintenance of the Hb Levels in CKD Patients on Dialysis , Treated According to Routine Clinical Practice
Brief Title: An Observational Study of Mircera (Methoxy Polyethylene Glycol-Epoetin Beta) in Chronic Kidney Disease Patients on Dialysis With Renal Anemia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25475
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the use in clinical practice and efficacy of Mircera (methoxy polyethylene glycol-epoetin beta) in chronic kidney disease patients on dialysis receiving Mircera for the treatment of chronic renal anemia. Eligible patients will be followed for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 65 years of age, inclusive
* Patients with chronic kidney disease on dialysis
* ESA naïve with Hb < 10 g/dL, or on treatment with ESAs other than Mircera and Hb within the target range of 10-12 g/dL
* Adequate irons status as judged by the treating physician

Exclusion Criteria:

* Hypersensitivity to recombinant human erythropoietin, polyethylene glycol or to any constituent of the study medication
* Clinically significant concomitant disease or disorder as defined by protocol
* Clinical suspicion of pure red cell aplasia (PRCA)
* Planned elective surgery during the study period , except for cataract surgery or vascular access surgery
* Transfusion of red blood cells in the previous 2 months
* Pregnant women
* Contraindications for Mircera according to local prescribing information or as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease on dialysis receiving treatment with Mircera for chronic renal anemia
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2011-04-30 (Actual); Primary Completion 2013-09-30 (Actual); Study Completion 2013-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- India (7):
  - Sir Gangaram Hospital, New Delhi, National Capital Territory of Delhi
  - Ahmedabad Dialysis Centre, Ahmedabad
  - Excel Center, Guwahati
  - ESIS Hospital; Department of Nephrology, Kolkata
  - Vertex Hospital, Mumbai
  - Apollo Indraprastha Hospitals; Nephrology, New Delhi
  - Aditya Birla Memorial Hospital, Pune

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 127 participants were enrolled from 7 centers in India. This study was conducted between 14 April 2011 and 23 September 2013.
Pre-assignment Details: Out of 127 participants enrolled in the study, 1 participant was enrolled wrongly and data for 2 participants were not available at the study Centre. Therefore, 124 participants were evaluated in this study.
Groups:
- C.E.R.A.: Participants with chronic renal anemia received C.E.R.A according to routine clinical practice treatment in line with approved prescribing information for a duration of 6 months/24 weeks.
Period: Overall Study
Arm/Group | C.E.R.A.
Started | 124
Completed | 102
Not Completed | 22
Not completed — Adverse Event | 1
Not completed — Death | 4
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 10
Not completed — Non-compliance by the participants | 3

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat (ITT) population included all the participants who received at least 1 dose of C.E.R.A and for whom data for at least one follow-up variable was available
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.1 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 83
Height [Mean (Standard Deviation); unit: Centimeters] — For mean height of participants n = 112 as height of some participants was not captured.
  Centimeters | 157.83 (10.056)

OUTCOME MEASURES:

1. Primary Outcome: Mean Age of Participants Treated With C.E.R.A
Description: Age was calculated on screening/Baseline visit day by using formula: Age = (Screening visit date - Date of birth)/365.25
Time Frame: Baseline (Week 0)
Population: The safety population included all participants enrolled into the study.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 124
Years | 48.1 (12.26)

2. Primary Outcome: Mean Weight of Participants Treated With C.E.R.A
Description: Weight of the participants was measured at the Baseline and summarized with descriptive statistics.
Time Frame: Baseline (Week 0)
Population: The safety population included all participants enrolled into the study. The analysis population reflects those participants whose weights were assessed at baseline.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 119
Kilograms | 57.44 (13.269)

3. Primary Outcome: Number of Participants With Co-morbidity Treated With C.E.R.A
Description: Co-morbidity is the presence of one or more additional disorders (or diseases) co-occurring with a primary disease or disorder; or the effect of such additional disorders or diseases. Co-morbid participants with renal and urinary disorders, vascular disorders, metabolism and nutrition disorders were reported.
Time Frame: Up to Week 24
Population: The safety population included all participants enrolled into the study.
Measure: Number; unit: Number of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 124
Number of participants
  Total comorbid participants | 107
  Comorbidity, renal and urinary disorders | 63
  Comorbidity, vascular disorders | 61
  Comorbidity, metabolism and nutrition disorders | 46

4. Primary Outcome: Mean Time Required to Achieve Target Hemoglobin Range
Description: The target range of hemoglobin (Hb) was 10-12 gram/deciliter (g/dL). Time to achieve target range = (Date of Hb evaluation when participant achieved target Hb range at first time - visit date of first dosing) + 1
Time Frame: Up to Week 24
Population: ITT population included all the participants who received at least 1 dose of C.E.R.A (Week 0) and for whom data for at least one follow-up variable was available. The analysis population reflects those participants whose Hb value was less than (<) 10 g/dL at enrollment.
Measure: Mean (Standard Deviation); unit: Week
Groups:
- C.E.R.A.: Participants with Hb less than (<) 10 g/dL at enrollment were evaluated for correction of anemia.
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 95
Week | 11.66 (5.652)

5. Primary Outcome: Percentage of Participants Achieved Target Range of Hemoglobin
Description: The target range of Hb was 10-12 gram/deciliter (g/dL). Time to achieve target range = (Date of Hb evaluation when participant achieved target Hb range at first time - visit date of first dosing) + 1. The percentage of participants with Hb < 10 g/dL at enrollment, achieving the target range of hemoglobin 10-12 g/dL was reported.
Time Frame: Up to Week 24
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 95
Percentage of participants | 74.7

6. Secondary Outcome: Number of Participants Achieving Hb Target Range (10-12 Hb g/dL) at Least Once During the Study
Description: For correction of anemia, number of participants achieving Hb target range (10-12 g/dL) at least once during the study were reported.
Time Frame: Up to Week 24
Population: ITT population included all the participants who received at least 1 dose of C.E.R.A (Week 0) and for whom data for at least one follow-up variable was available.
Measure: Number; unit: Number of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 121
Number of participants | 83

7. Secondary Outcome: Mean Time Spent by Participants in the Hb Target Range
Description: Maintenance of target Hb was evaluated by assessing the mean time spent by participants in target Hb range. The target Hb range in the study was 10-12 g/dL.
Time Frame: Up to Week 24
Population: ITT population included the participants who received at least 1 dose of C.E.R.A (Week 0) and for whom data for at least one follow-up variable was available.
Measure: Mean (Standard Deviation); unit: Week
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 121
Week | 13.54 (6.143)

8. Secondary Outcome: Evaluation of Route of Administration for C.E.R.A
Description: C.E.R.A. was administered by Intravenous (IV) and Subcutaneous (SC) route of administration. The frequency (number of injections) for both of these routes of administration used in the study was reported.
Time Frame: Up to Week 24
Population: The safety population included all participants enrolled into the study
Measure: Number; unit: Number of injections
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 124
Number of injections
  Intravenous administration | 11
  Subcutaneous administration | 647

9. Secondary Outcome: Evaluation of Dose Per Injection of C.E.R.A
Description: The dosing and titration of C.E.R.A treatment were at the discretion of the investigator in accordance with local clinical practice or approved prescribing information. Mean dose per injection of C.E.R.A received by participants was reported.
Time Frame: Up to Week 24
Population: The safety population included all participants enrolled into the study
Measure: Mean (Standard Deviation); unit: Microgram
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 124
Microgram | 64.0 (21.30)

10. Secondary Outcome: Number of Participants Received Concomitant Medications
Description: Medications that were used during the study treatment period (from the first dose date of study medication to the end of the study) were included as concomitant medications. The prescribed concomitant medications (in greater than or equal to 10% of participants) in the study were prazosin, torasemide, vitamin and nutritional supplements, omeprazole, amlodipine, calcium supplements, calcitriol, and clonidine. Participants treated with the each of these concomitant medications were reported.
Time Frame: Up to Week 24
Population: The safety population included all participants enrolled into the study
Measure: Number; unit: Number of participants
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 124
Number of participants | 122

11. Primary Outcome: Percentage of Participants Who Had Received Treatment With Other Erythropoiesis-Stimulating Agents Maintaining Hb Level Within 1 Gram/Deciliter of Baseline Value During Study Period in Participants.
Description: Percentage of participants maintaining Hb level within 1 g/dL of baseline value during study period who had received treatment with other Erythropoiesis-Stimulating Agents (ESAs) were reported.
Time Frame: Up to Week 24
Population: ITT population included all the participants who received at least 1 dose of C.E.R.A (Week 0) and for whom data for at least one follow-up variable was available. The analysis population reflects those participants who had been on other ESAs and had Hb greater than or equal to (≥)10 g/dL at baseline.
Measure: Number; unit: Percentage of participants
Groups:
- C.E.R.A.: Participants with chronic renal anemia who had been on other ESAs and had Hb greater than or equal to (≥)10 g/dL at baseline.
Arm/Group | C.E.R.A.
Number analyzed (Participants) | 25
Percentage of participants | 20

ADVERSE EVENTS:
Time Frame: Up to Week 24
Description: An Adverse Event is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | C.E.R.A.
Serious Adverse Events (participants affected / at risk) | 6/124
Other Adverse Events (participants affected / at risk) | 21/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=124)
Peritonitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1 — General Disorders And Administrations
Death (General disorders) | 2 — General Disorders And Administrations
Pneumonia (Infections and infestations) | 1
Chronic renal failure (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C.E.R.A. (N=124)
Peritonitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 4 — General Disorders And Administrations
Pyrexia (General disorders) | 7 — General Disorders And Administrations
Cough (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.